CLINICAL TRIAL: NCT02899520
Title: Evaluation of Programs of Reeducation for Urinary Incontinence in Woman
Acronym: ReedPerinee
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in the clinical practices
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014/09; 2014-A00709-38 (Other: ANSM)
Record Dates: First submitted 2016-09-09; First posted 2016-09-14 (Estimated); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Active Comparator): Reference method
  Interventions: Other: Reference method
- Group B (Experimental): CMP ® method (Knowledge and Control of Perineum)
  Interventions: Other: CMP ® method

INTERVENTIONS:
Other: Reference method — Electrostimulation associated to perineal training
  Arms: Group A
Other: CMP ® method — Method based on Knowledge and Control of Perineum
  Arms: Group B

SUMMARY:
The objective of this study is to compare two methods of pelvic floor muscle training: reference method versus CMP ® method ( (Connaissance et Maîtrise de Périnée : Knowledge and Control of Perineum)

ELIGIBILITY:
Inclusion Criteria:

* Patients more than 18 years old and less than 75 years
* Patients presenting an urinary incontinence of effort or mixed symptomatic associated with a pelvic statics disorder
* Patients with a perineale reeducation prescription
* Patients affiliated to a national insurance scheme or benefiting from such a program
* Patients having given her written consent form

Exclusion Criteria:

* Nulliparous woman
* Patients already operated for their incontinence
* Patients with a prolapse of higher level at the stage II of the classification POP-Q (Pelvic Organ Prolapse Quantification)
* Pregnant women
* Patients presenting an associated anal incontinence,
* Patients presenting a cancellation (section of marrow, syringomyelia for example) or an inversion of perineum control
* Patients having given birth less than 6 months before the care
* Patients having benefited from a pelvi-périnéale reeducation in the previous 12 months,
* Patients presenting psychiatric disease
* Patients presenting a vaginismus,
* Patients presenting a contraindication to the practice of the electrostimulation.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-11-10 (Actual); Primary Completion 2019-10-18 (Actual); Study Completion 2019-10-18 (Actual)

PRIMARY OUTCOMES:
USP (Urinary Symptoms Profile) score | 38 weeks
  Urinary Symptoms Profile score

CONTACTS AND LOCATIONS:
Overall Officials: Sophie FLANDIN-CRETINON, Principal Investigator — Hopital Foch
Locations (1):
- Hopital Foch, Suresnes, France